CLINICAL TRIAL: NCT03447847
Title: Effect of Composition and Timing of Ingestion of Fluids on the Urinary Excretion of Lithogenic Substances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pietro Manuel Ferraro, Assistant Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 43111/16
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Healthy
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 (Experimental): A=oligomineral water, B=oligomineral water
  Interventions: Other: Water
- Phase 2 (Experimental): A=oligomineral water, B=bicarbonate-rich water
  Interventions: Other: Water
- Phase 3 (Experimental): A=bicarbonate-rich water, B=oligomineral water
  Interventions: Other: Water
- Phase 4 (Experimental): A=bicarbonate-rich water, B=bicarbonate-rich water
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — 1 liter of water in meals; 1 liter out of meals

SUMMARY:
Interventional crossover study on healthy volunteers aimed at evaluating the effect of the composition and timing of ingestion of different types of water on the urinary excretion of lithogenic substances; the study will also analyze the effect of potassium citrate on urine pH and lithogenic substances

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years

Exclusion Criteria:

* Chronic malabsorption
* Recurrent urinary tract infections
* History of kidney stones

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Urine composition | Assessed the same day of water ingestion

CONTACTS AND LOCATIONS:
Locations (1):
- Divisione di Nefrologia, Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferraro PM, Baccaro R, Baroni S, D'Alessandri L, Carpenito C, Di Daniele N, Urbani A, Gambaro G. Effect of water composition and timing of ingestion on urinary lithogenic profile in healthy volunteers: a randomized crossover trial. J Nephrol. 2021 Jun;34(3):875-881. doi: 10.1007/s40620-020-00769-2. Epub 2020 Jun 8. PMID 32514990